CLINICAL TRIAL: NCT01000792
Title: 3-D Visualization of the Anti-Obstructive Effect of Levocetirizine - A Monocentric Clinical Trail With One Patient (Phase-IV-Study)
Brief Title: 3-D Visualization of the Anti-Obstructive Effect of Levocetirizine
Acronym: LevoNasalFlo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clinical Research International Limited (Industry)
Responsible Party: Prof. Dr. med. Dipl.-Ing. Ralph Mösges, CRI - Clinical Research International Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRI-2009-09-001-IV
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — levocetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levocetirizine (Experimental): Levo 5 mg o.d.
  Interventions: Drug: Levocetirizine

INTERVENTIONS:
Drug: Levocetirizine — The study drug is Xyzal® 5 mg (API: levocetirizine dihydrochloride). 28 film tablets will be dispensed. Oral intake should be performed once daily (administration in the evening).
Drug: Levocetirizine — Levocetirizine

SUMMARY:
The prevalence of allergic rhinitis is high and appears to be rising worldwide. Therefore, it is important and necessary to understand and visualize therapy effects on this disease. In this study we will demonstrate the effect of levocetirizine on nasal cavity dimensions by assessing not only standard nasal flow diagnostics such as rhinomanometry and acoustic rhinometry, but supplement exami¬nation procedures with long-term rhinometry and magnetic resonance imaging (MRI). With the aid of a virtual model and computer fluid dynamics, we are able to simulate nasal air flow and provide three-dimensional visualization of the computed flow.

In previous trials ([Bachert], [deBlic], [Day] and [Deruaz]) it has been shown that allergic symptoms, especially nasal congestion, diminish significantly under treatment with levocetirizine. We will demonstrate this anti-obstructive effect by comparing the reaction to nasal allergen challenge before and after four-week treatment with levocetirizine.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be informed and give written informed consent for study participation
* Subject must be able to adhere to dose and visit schedules and meet study requirements
* Subject must be aged 18 to 65 (inclusive); gender and race are irrelevant
* Subject must have at least a two-year history of allergic rhinitis consistent with persistent allergic rhinitis (defined as symptoms of allergic rhinitis present on four days or more per week or for four or more consecutive weeks per year)
* In the previous pollen season, subject must have been sufficiently symptomatic, with a T6SS (reflective) symptoms severity score of at least 10 (out of max. 18). (Symptoms include nasal itching, sneezing, rhinorrhea, congestion, conjunctival itching, redness and tearing graded on a scale of 0 -absent, 1 - mild, 2 - moderate, 3 - severe)
* Subject must have a positive skin prick test at screening to one or more allergens in the local panel of seasonal allergens (e.g. grass, tree pollen), but not to perennial allergens. Subject must demonstrate an antigen-induced skin prick wheal of at least 3mm greater in diameter than the diluent control.
* Subject must have had a positive nasal allergen challenge within the previous six months. (see [Riechelmann])
* Nonsterile or premenopausal female subjects must use a medically accepted method of birth control, e.g. oral contraceptives

Exclusion Criteria:

* Failure to fulfill all of the above mentioned inclusion criteria
* Insufficient ability to understand the nature, scope and possible consequences of the study
* Insufficient legal competence or insufficient knowledge of the German language
* Participation in another clinical trial within the previous three months
* Pregnancy or lactation
* Positive skin prick test to frequently occurring perennial allergens, e.g. house dust mites, cats
* History of anaphylaxis and/or severe local reactions to skin testing with allergens
* Intolerable symptoms that would make participating in the study unbearable, especially the 45 min MRI-session
* Any viral inflammation of the upper respiratory system, acute or chronic sinusitis, rhinitis medicamentosa, nasal polyps, clinically relevant anatomic deviations of the nose, active or inactive tuberculosis of the respiratory tract, or asthma other than mild intermittent asthma treated with ß2-agonists on an as-needed basis
* Any kind of clinically significant disease, especially any signs of active persistent allergic rhinitis, which would interfere with the study evaluations.
* Known intolerance to levocetirizine or any other components of the study drugs
* Surgery of the nose or the nasal sinuses within the previous six months
* Any deviation from the norm in the physical investigation of any disease which in the investigator's judgment might require impermissible medication, influence study performance and results or affect the patients safety
* Intake of drugs which might interfere with the study results
* History of alcohol or drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-11; Primary Completion 2010-01 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Improvement of nasal flow | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Mösges, M.D., Principal Investigator — CRI-Ltd
Locations (1):
- HNO-Praxis Dr. Pasch/Prof. Schlöndorff, Aachen, North Rhine-Westphalia, Germany